CLINICAL TRIAL: NCT00444379
Title: A Randomized Comparison of Protease Inhibitor-based Versus Non-nucleoside Reverse Transcriptase Inhibitor-based Antiretroviral Therapy for Initial Treatment of Individuals With AIDS-related Kaposi's Sarcoma in Sub-Saharan Africa
Brief Title: Anti-Retrovirals for Kaposi's Sarcoma
Acronym: ARKS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Gilead Sciences (Industry); Abbott (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIH/NCI Grant #: R01 CA119903
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Kaposi's Sarcoma; HIV Infections
Keywords: Kaposi's sarcoma; KSHV; AIDS; HHV-8; treatment naive
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Lopinavir; Ritonavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PI-based HAART regimen (Active Comparator): PI-based HAART regimen (lopinavir/ritonavir plus emtricitabine/tenofovir)
  Interventions: Drug: Lopinavir/ritonavir plus Emtricitabine/Tenofovir versus Efavirenz plus Emtricitabine/Tenofovir
- non-nucleoside reverse transcriptase inhibitor (Active Comparator): non-nucleoside reverse transcriptase inhibitor (NNRTI)-based HAART regimen (efavirenz plus emtricitabine/tenofovir)
  Interventions: Drug: Lopinavir/ritonavir plus Emtricitabine/Tenofovir versus Efavirenz plus Emtricitabine/Tenofovir

INTERVENTIONS:
Drug: Lopinavir/ritonavir plus Emtricitabine/Tenofovir versus Efavirenz plus Emtricitabine/Tenofovir — Lopinavir/ritonavir 200/50mg plus Emtricitabine/Tenofovir 200/300mg versus Efavirenz 600mg plus Emtricitabine/Tenofovir 200/300mg
  Other Names: Lopinavir/ritonavir Aluvia (ALUABT); Efavirenz Stocrin (EFVBMM); Emtricitabine/Tenofovir Truvada (TRUGLD)

SUMMARY:
The primary purpose of this study is to determine whether a protease inhibitor-based antiretroviral regimen is more efficacious than a non-nucleoside reverse transcriptase inhibitor-based antiretroviral regimen in promoting the regression of KS tumor burden in persons with AIDS-related KS in Africa.

DETAILED DESCRIPTION:
With the advent of the HIV epidemic, Kaposi's sarcoma (KS) is now the most common adult cancer in many parts of sub-Saharan Africa. In HIV-infected patients with KS in developed settings, the initiation of highly active anti-retroviral therapy (HAART) has been associated with regression of the tumor, in many but not all cases, even in the absence of conventional chemotherapy. However, it is not known which specific antiretroviral drugs or regimens are critical to convey HAART's anti-KS effect. In particular, it is not known whether the anti-KS effects of protease inhibitors (PI) in vitro and in animal models translate into improved clinical outcomes as compared to non-PI-based HAART regimens. To address this, we will determine whether a PI-based HAART regimen (lopinavir/ritonavir plus emtricitabine/tenofovir) is superior to a non-nucleoside reverse transcriptase inhibitor (NNRTI)-based HAART regimen (efavirenz plus emtricitabine/tenofovir) in promoting the regression of KS tumor burden in persons with AIDS-related KS in sub-Saharan Africa. We will enroll 224 patients with AIDS-related KS in Kampala, Uganda, randomly assign them to either a PI-based HAART or an NNRTI-based HAART regimen, and observe them for one year to determine the response in their KS to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* HIV-1 infection
* No prior antiretroviral therapy of any duration, including prior use to prevent perinatal transmission within prior six months.
* No prior chemotherapy or radiotherapy for KS
* Presence of Kaposi's sarcoma, documented by biopsy by the Pathology Department at Mulago Hospital, with at least one mucocutaneous lesion (including oral or genital mucosal lesions), each at least 0.6 x 0.6 cm in perpendicular diameters.
* Laboratory values obtained within 21 days prior to randomization: absolute neutrophil count equal to or more than 1000/mm3; hemoglobin > 9.0 g/dL; platelet count > 50,000/mm3; creatinine < 2 times upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 times ULN; and alkaline phosphatase and total bilirubin < 2 times ULN.
* In women, negative urine pregnancy test within 28 days of randomization and just before randomization.
* If a woman of child-bearing potential (i.e., not yet reached menopause or undergone hysterectomy, bilateral oophorectomy, or tubal ligation), must be willing to use at least two of the following methods of contraception, to be provided by the study: condoms (male or female), IUD, or hormone-based therapy, e.g., contraceptive pills, Norplant or Depo-Provera.
* Candidate currently resides within Uganda and does not intend to relocate away from current geographical area of residence for the duration of study participation.
* Karnofsky performance score of 70 or more

Exclusion Criteria:

* Extensive degree of mucocutaneous KS, which would typically require chemotherapy or radiotherapy. This is defined by any of the following:

  * One or more bulky cutaneous lesions, defined as at least 5.0 cm in greatest diameter across the surface of the skin and at least 3 cm in height
  * One or more mucocutaneous lesions exhibiting ulceration
  * One or more oral lesions that interfere with swallowing
* Suggestion of pulmonary or gastrointestinal visceral KS, as evidenced by any of the following:

  * Abnormal chest x-ray within 21 days prior to randomization which is otherwise unexplained, unless the x-ray is unchanged compared with at least 60 days earlier
  * Positive occult blood stool testing within 21 days prior to randomization or history of overt bleeding from the mouth or rectum in the 21 days prior to randomization
* Facial lymphedema or lymphedema in any other body region which causes symptoms (e.g., pain) or functional disability (e.g., any less than 85% active range of motion in a large joint)
* Evidence of currently active, untreated opportunistic infection or malignancy (not including Kaposi's sarcoma); or unexplained temperature which is > 38.5 degrees C
* Use of drugs, within the prior 28 days, contraindicated while taking lopinavir/ritonavir or efavirenz because of effects on the cytochrome P450 system. These include propafenone, astemizole, terfenadine, rifampin, rifapentine, ergot derivatives, cisapride, lovastatin, simvastatin, pimozide, midazolam, and triazolam.
* Active drug or alcohol use that, in the investigators' opinion, would interfere with study participation
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2007-04; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Blinded assessment of the change in the burden of KS lesions
  survival

SECONDARY OUTCOMES:
CD4+ T cell count and HIV plasma HIV RNA levels
KSHV DNA levels in saliva and blood
Humoral and cellular KSHV immune response markers
Quality-of-life assessment
Incidence of Kaposi's sarcoma-associated Immune Reconstitution Inflammatory Syndrome (KS-IRIS)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jeffrey N Martin, MD, MPH, Principal Investigator — University of California, San Francisco; Dr. Edward K Mbidde, MBChB, MMed, Principal Investigator — MRC/UVRI and LSHTM Uganda Research Unit
Locations (1):
- Infectious Diseases Institute, Mulago Hospital, Kampala, Uganda

REFERENCES:
- See also: Medline Plus- Health Information — http://www.nlm.nih.gov/medlineplus/kaposissarcoma.html